CLINICAL TRIAL: NCT01038414
Title: Duration of Behavioral Counseling Treatment Needed to Optimize Smoking Abstinence
Acronym: EDC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harvard University Faculty of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Arthur J. Garvey, Ph.D., Harvard School of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01DA12165-8; 5R01DA012165 (NIH)
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Tobacco Addiction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Brief-Duration Counseling (Placebo Comparator): 3-Month Duration
  Interventions: Behavioral: Extended Duration Behavioral Smoking Cessation Counseling
- Moderate Duration Counseling (Active Comparator): 6-Month Duration
  Interventions: Behavioral: Extended Duration Behavioral Smoking Cessation Counseling
- Extended Duration Counseling (Active Comparator): 12-Month Duration
  Interventions: Behavioral: Extended Duration Behavioral Smoking Cessation Counseling

INTERVENTIONS:
Behavioral: Extended Duration Behavioral Smoking Cessation Counseling — Subjects are randomized to one of 3 behavioral treatments: (1) Brief Duration (3 month) smoking-cessation counseling; (2) Moderate Duration (6 month) counseling; or (3) Extended Duration (12 month) counseling
  Other Names: Extended-Duration Behvioral Smoking-Cessation Counseling

SUMMARY:
The purpose of this study is to determine if extending the behavioral smoking-cessation treatment period to one year will significantly improve cessation outcomes among those planning a quit attempt.

ELIGIBILITY:
Inclusion Criteria:

* Daily Cigarette Smokers

Exclusion Criteria:

* Smokers with active atherosclerotic heart disease, severe cardiac arrhythmias, uncontrolled hypertension, severe peripheral vascular disease, pre-controlled diabetes mellitus, pregnancy, lactation or likely to become pregnant during the study period, and chronic dermatologic disease.
* Smokers who meet DSM-IV lifetime criteria for conditions such as schizo-affective disorder and schizophrenia, bi-polar disorder, or who have had alcohol or drug dependence issues within the past year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2008-02; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects abstinent by treatment group at 1 year post-cessation. | One year

SECONDARY OUTCOMES:
Proportion of subjects abstinent by treatment group at 2 years post-cessation. | Two years

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard School of Dental Medicine, Boston, Massachusetts, United States